CLINICAL TRIAL: NCT05600530
Title: Validity and Reproducibility of A Self-administered Web-based 24-hour Dietary Assessment Tool Among Danish Adults Against Objective Measures
Brief Title: Validity and Reproducibility of Dietary Assessment Against Objective Measures
Acronym: VALID
Status: Completed | Type: Observational
Sponsor: Inge Tetens (Other)
Responsible Party: Sponsor-Investigator, Inge Tetens, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: M243
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Validation Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine and blood samples to measure biomarker excretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study with repeated measurements among healthy Danish adults to assess the validity and reproducibility of a self-administered 7-day web-based dietary assessment tool, myfood24® tested against objective biomarkers.

DETAILED DESCRIPTION:
Healthy volunteers (age 35-70 yrs; BMI 22-32) will be recruited for the study. Informed consent will be obtained and participants will complete a self-administered web-based 7-day 24-hour dietary recall tool (myfood24®).Validity of this dietary registration tool will be assessed by comparing the estimated intake of selected nutrients (protein, energy) and selected food groups (fruit and vegetables, whole grain, coffee, alcoholic beverages) against objective biomarkers obtained from a 24-hour urine sample, through a measurement of resting energy metabolic rate, and from a fasting blood sample, respectively. Reproducibility will be assessed by comparison of the results from two self-administered web-based 7-day 24-hour dietary recalls obtained 4 weeks (± 1 weeks) apart.

ELIGIBILITY:
Inclusion criteria:

* Apparently healthy adults between 35 and 70 years old
* Body mass index (BMI) between 22-32 kg/m2
* Weight stable defined as gain or loss of < 2.5% body weight during the past 3 months;
* Willingness to maintain current dietary and physical activity habits throughout the study period.
* Have high-speed internet access;
* Able to speak, read and write Danish;
* Willing to visit the Department of Nutrition, Exercise, and Sports (NEXS).

Exclusion Criteria:

* Clinically diagnosed chronic disease,
* use of corticosteroids or other medication that would potentially affect the nutrient metabolism or excretion of biomarkers of interest,
* presence of food allergy or intolerance that requires a special diet,
* pregnancy and lactation,
* excess physical activity (>5h/week of high intensity),
* current participation in another trial

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Danish adults
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Validation of protein intake | 7 days
  Agreement between mean protein intake per day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and nitrogen excretion in a 24-hr urine sample (urea corrected for creatine).

SECONDARY OUTCOMES:
Validation of energy intake | 7 days
  Agreement between mean energy intake per day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and resting metabolic rate (measured by ventilated hood).
Validation of vegetable and fruit intake | 7 days
  Agreement between mean intake of vegetable and fruit per day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and concentration of folate in a fasting blood sample.
Validation of whole grain intake | 7 days
  Agreement between intake of whole grain per day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and excretion of alkylresorcinols in a fasting blood sample.
Validation of alcohol intake | 7 days
  Agreement between mean alcohol intake pr day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and excretion of ethanol and ethyl conjugates in a 24-hr urine sample.
Validation of coffee intake | 7 days
  Agreement between mean coffee intake per day assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) and excretion of trigonelline and cyclo(isoleucylprolyl) in a 24-hr urine sample.
Reproducibility of dietary registration | Two times 4 weeks (+/- 1 week) apart
  Agreement between two dietary intake measurements assessed by the self-administered 7-day web-based dietary assessment tool (myfood24) obtained 4 (± 1 week) apart.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Tetens, PhD, Principal Investigator — Professor
Locations (1):
- University of Copenhagen, Frederiksberg, DK, Denmark

IPD SHARING:
Plan to Share IPD: Undecided